CLINICAL TRIAL: NCT05532917
Title: Impact of 2014 ACC/AHA Perioperative Guidelines on Cardiological Resource Use in Noncardiac Surgery Patients
Brief Title: Cardiology Consultation in Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Atar, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: 10.1.2022 128/21
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Infarction; Surgery-Complications
Keywords: ACC/AHA guidelines; Perioperative cardiac risk; Cardiology consultation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gupta group: Cardiology consultation requested using Gupta score
  Interventions: Other: Gupta score
- Non-Gupta group: Number of cardiology consultations requested without using Gupta score

INTERVENTIONS:
Other: Gupta score — The Gupta score is presented as an interactive risk calculation program in the 2014 guideline of the ACC/AHA. The Gupta score developed with this MICA model identified five predictors of perioperative myocardial infarction and cardiac arrest: type of surgery, functional status, creatinine increase (>130 mmol/L or >1.5 mg/dL), age, and American Association of Anesthesiologists (ASA) class. The frequency of cardiology consultation requests will be investigated according to the use of the Gupta score.
  Groups: Gupta group

SUMMARY:
Recently, a predictive model has been developed to assess the risk of myocardial infarction or cardiac arrest (MICA) during and after surgery using the American Society of Surgeons' National Surgical Quality Improvement Program (NSQIP) database. In this MICA model, 180 hospital databases were used in 2007 and 2008 and included more than 200 000 patients. The Gupta score developed with this MICA model identified five predictors of perioperative myocardial infarction and cardiac arrest: type of surgery, functional status, creatinine increase (>130 mmol/L or >1.5 mg/dL), age, and American Association of Anesthesiologists (ASA) class. The Gupta score is presented as an interactive risk calculation program in the 2014 guideline of the ACC/AHA. The risk can be calculated simply and accurately at the bedside or clinic. The Gupta score is in spreadsheet format and can be downloaded online at http://www.surgicalriskcalculator.com/miorcardiacarrest. Unlike the previously used indexes, a scoring system has not been established. An estimate of the probability of myocardial infarction/cardiac arrest is provided for individual patients.

In this study, the primary aim was to compare the frequency of cardiology consultation requests according to the use of the Gupta score. The secondary aim is to evaluate the perioperative clinical results (coronary angiography, ECHO, acute coronary syndrome, arrhythmia, 30-day mortality, etc.).SPSS 21.0 (Version 22.0, SPSS, Inc, Chicago, IL, USA) program will be used for statistical analysis. After applying the Shapiro-Wilk test for normality, the student's t-test will be used if the distribution is normal, and the Mann-Whitey U test will be used if the distribution is not normal. Fisher's exact test or chi-square test will be used for categorical variables. Results p<0.05 will be considered significant.

DETAILED DESCRIPTION:
All patients undergoing non-cardiac surgery are at risk of major perioperative cardiovascular events. Cardiac complications account for 42% of the overall complications of these surgeries. Therefore, cardiologists are the most frequently consulted specialists in preoperative evaluation. Unnecessary cardiology consultations may cause comments that will not affect the practice of anesthesia, inappropriate tests and interventions, and delay in the surgical procedure.

Recently, a predictive model has been developed to assess the risk of myocardial infarction or cardiac arrest (MICA) during and after surgery using the American Society of Surgeons' National Surgical Quality Improvement Program (NSQIP) database. In this MICA model, 180 hospital databases were used in 2007 and 2008 and included more than 200 000 patients. The Gupta score developed with this MICA model identified five predictors of perioperative myocardial infarction and cardiac arrest: type of surgery, functional status, creatinine increase (>130 mmol/L or >1.5 mg/dL), age, and American Association of Anesthesiologists (ASA) class. The Gupta score is presented as an interactive risk calculation program in the 2014 guideline of the ACC/AHA. The risk can be calculated simply and accurately at the bedside or clinic. The Gupta score is in spreadsheet format and can be downloaded online at http://www.surgicalriskcalculator.com/miorcardiacarrest. Unlike the previously used indexes, a scoring system has not been established. An estimate of the probability of myocardial infarction/cardiac arrest is provided for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-cardiovascular surgery
* Patients evaluated routinely preoperatively in the anesthesiologist preoperative outpatient clinic

Exclusion Criteria:

* Emergency surgeries
* ASA Physical Status V
* Patients undergoing cardiovascular surgery
* Minor surgeries
* Patients who did not want to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who will be referred to the anesthesia polyclinic and will undergo non-cardiac surgery will be included in the study. Cardiology consultation will be requested from these patients according to the Gupta score. Additional tests or examinations may be requested if the cardiologist deems it necessary.
Sampling Method: Probability Sample
Enrollment: 898 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Gupta score | perioperative period
  The frequency of cardiology consultation requests will be compared according to the use of the Gupta score.

SECONDARY OUTCOMES:
Perioperative clinical results | perioperative period
  Perioperative clinical results (coronary angiography, ECHO, acute coronary syndrome, arrhythmia, 30-day mortality, etc.) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Science, Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cinello M, Nucifora G, Bertolissi M, Badano LP, Fresco C, Gonano N, Fioretti PM. American College of Cardiology/American Heart Association perioperative assessment guidelines for noncardiac surgery reduces cardiologic resource utilization preserving a favourable clinical outcome. J Cardiovasc Med (Hagerstown). 2007 Nov;8(11):882-8. doi: 10.2459/JCM.0b013e3280122d63. PMID 17906472
- [Background] Glance LG, Faden E, Dutton RP, Lustik SJ, Li Y, Eaton MP, Dick AW. Impact of the Choice of Risk Model for Identifying Low-risk Patients Using the 2014 American College of Cardiology/American Heart Association Perioperative Guidelines. Anesthesiology. 2018 Nov;129(5):889-900. doi: 10.1097/ALN.0000000000002341. PMID 30001221
- [Background] Madi-Jebara S, Chalhoub V, Jabbour K, Yazigi A, Haddad F, Richa F, El-Hage C, Yazbeck P. [Audit on preoperative cardiac evaluation before non-cardiac surgery: the importance of a pocket guide to improve the anaesthesist's adhesion to ACC/AHA guidelines]. Ann Fr Anesth Reanim. 2009 Oct;28(10):850-4. doi: 10.1016/j.annfar.2009.08.007. Epub 2009 Oct 29. French. PMID 19879104